CLINICAL TRIAL: NCT04719845
Title: Dilatation Versus Endoscopic Laser Resection in Simple Benign Tracheal Stenosis : a Randomized Controlled Trial
Brief Title: DilAtation Versus Endoscopic Laser Resection in Simple Benign trAcheal sTEnosis
Acronym: AERATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Marc Fortin, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-3573
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Tracheal Stenosis
MeSH Terms: conditions — Tracheal Stenosis | interventions — Dilatation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic laser resection (Experimental): Using CO2, diode or similar wavelenght laser the stenotic tracheal segment will be vaporized allowing a less than 20% residual stenosis. Dilatation will not be performed after laser resection for residual stenosis.
  Interventions: Procedure: Endoscopic laser resection
- Dilatation (Experimental): Using a ballon or rigid bronchoscope the stenotic tracheal segment will be dilated with or without previous radial incision with electrocautery or laser.
  Interventions: Procedure: Dilatation

INTERVENTIONS:
Procedure: Endoscopic laser resection — Laser resection
  Arms: Endoscopic laser resection
Procedure: Dilatation — Dilatation
  Arms: Dilatation

SUMMARY:
Multicenter randomized controlled trial comparing endoscopic laser resection vs dilatation in benign tracheal stenosis.

DETAILED DESCRIPTION:
An observational study suggests the superiority of endoscopic laser resection over dilatation in idiopathic tracheal stenosis but little litterature has been published on the subject. Hence we decided to design a prospective multicenter open label randomized controlled trial to compare the two interventions. Patients refered for endoscopic treatment of a simple benign tracheal stenosis will be randomized to endoscopic laser resection or dilatation. Randomisation will be stratified for center, type of stenosis (idiopathic vs other) and history of previous endoscopic treatment. Patients will be blinded to treatment but not physician. All patients will be treated with proton pump inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Benign simple tracheal stenosis (length of stenosis <1cm without underlying cartilage damage) with planned endoscopic treatment (first treatment or recurrence)

Exclusion Criteria:

* Less than 18 years old
* Pregnant
* Incapacity to give informed consent
* Underlying inflammatory suspected to be the cause of stenosis (ex : granulomatosis with polyangitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Relapse rate at 2 years of symptomatic tracheal stenosis (> 40%) requiring a new procedure | Within 2 years

SECONDARY OUTCOMES:
Relapse rate at 1 year of symptomatic tracheal stenosis (> 40%) requiring a new procedure | 1 year
Time to first symptomatic relapse of tracheal stenosis | 2 years
mMRC | 2 years
VAS | 2 years
Clinical COPD questionnaire | 2 years
VHI-10 | 2 years
SF-12 | 2 years
Measurement of stenosis by cephalo-caudal length at endoscopic follow-up at 1 year | Within 2 years
Rate of surgical resection following symptomatic recurrence | 2 years
Rate and type of complications and adverse effects depending on the procedure | 2 years

OTHER OUTCOMES:
Relapse rate at 2 years of symptomatic tracheal stenosis (> 40%) requiring a new procedure in the idiopathic and non idiopathic subroup as well as in the first episode and recurrence subgroups | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fortin, Principal Investigator — Fondation IUCPQ
Locations (4):
- Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Canada
- France (3):
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Hôpital Nord, Marseille
  - Hôpital Larrey, University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soumagne T, Guibert N, Atallah I, Lacasse Y, Dutau H, Fortin M. Dilation versus laser resection in subglottic stenosis: protocol for a prospective international multicentre randomised controlled trial (AERATE trial). BMJ Open. 2022 Mar 17;12(3):e053730. doi: 10.1136/bmjopen-2021-053730. PMID 35301206